CLINICAL TRIAL: NCT00136006
Title: The Burden of Chronic Obstructive Lung Disease (BOLD) Study
Brief Title: The Vancouver-BOLD Study: The Burden of Chronic Obstructive Lung Disease
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: P05-0061; 05-0965
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2013-01

CONDITIONS: Chronic Obstructive Lung Disease
Keywords: Epidemiology; Lung health; lung function; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Behavioral: Study to determine the burden of disease

SUMMARY:
This is a study of the lung health of the population of Vancouver and the extent of, and the risk factors for, chronic obstructive lung disease.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age and older
* Both sexes
* Random sample of population

Exclusion Criteria:

* Contraindication for lung function testing and serious life threatening illness.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of Vancouver, BC, Canada
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2005-08-01; Primary Completion 2013-12-01 (Actual); Study Completion 2013-12-01 (Actual)

PRIMARY OUTCOMES:
Lung health | 10 years
  Lung health of the population of Vancouver and the extent of, and the risk factors for, chronic obstructive lung disease

CONTACTS AND LOCATIONS:
Overall Officials: Wen Wang, Study Director — University of British Columbia
Locations (1):
- St.Paul's Hospital/Providence Health Care, Vancouver, British Columbia, Canada